CLINICAL TRIAL: NCT07051382
Title: Transcranial Sonographic Evaluation of Preterm Neonates Presenting With Seizures and Its Association With Intracranial Abnormalities
Brief Title: Transcranial Sonographic Evaluation of Preterm Neonates Presenting With Seizures and Its Association With IA
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/921
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Intracranial Abscess

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transcranial Sonographic Examination (Cranial Ultrasound) — No evidence of intracranial abnormalities such as intraventricular hemorrhage, germinal matrix hemorrhage, periventricular leukomalacia, hydrocephalus, or infarction.
  Brain structures were assessed to be age-appropriate for gestational development.

SUMMARY:
This study aimed to evaluate preterm neonates presenting with seizures using transcranial sonography (cranial ultrasound) to detect intracranial abnormalities.

DETAILED DESCRIPTION:
To determine the prevalence and types of intracranial abnormalities detected by transcranial sonography in preterm neonates who present with seizures, and to analyze the association between these findings and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Both genders during neonatal period i.e. up to 28 days of postnatal life.
* Seizures having any birth weight and gestational age.3.6.2

Exclusion Criteria:

* Preterm with Congenital spinal anomalies causing seizures such as spina-bifida, scoliosisetc.
* Extra-cranial anomalies causing seizures such as arteriovenous malformation (AVM) or metabolic diseases.

Ages: 1 Week to 20 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This group consisted of preterm neonates who presented with seizures and showed abnormalities on cranial ultrasound, such as: Germinal Matrix ,Hemorrhage (GMH) Intraventricular, Periventricular Leukomalacia (PVL) , Hydrocephalus , Cerebral infarction or parenchymal lesions.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Self Administred Questioner | 12 Months
  Self Administred Questioner for taking the data and values

CONTACTS AND LOCATIONS:
Locations (1):
- Mohmand medical complex hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan